CLINICAL TRIAL: NCT04587258
Title: Improving Cancer Screening and Prevention During the COVID-19 Pandemic in Underserved Populations of Rhode Island: A Community Based Quality Improvement Project of the Lifespan Cancer Institute
Brief Title: Improving Cancer Screening and Prevention During the COVID-19 Pandemic in Underserved Populations of Rhode Island
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: Blackstone Valley Community Health Care (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1613494-3
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Colorectal Cancer; Covid19
Keywords: Cancer screening; COVID19; Underserved communities; Community based-participation; Social Media; Informational videos; Facebook; Instagram; TikTok; Lifespan; Blackstone Valley; Central Falls; Pawtucket; Providence; Minorities; Equitable healthcare
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer: Subjects will be encouraged through informational videos and social media campaigns to visit their doctors to get screened for breast cancer using mammograms.
  Interventions: Behavioral: Informational videos and social media campaigns encouraging cancer screening.
- Colorectal Cancer: Subjects will be encouraged through informational videos and social media campaigns to visit their doctors to get screened for breast cancer using colonoscopies
  Interventions: Behavioral: Informational videos and social media campaigns encouraging cancer screening.

INTERVENTIONS:
Behavioral: Informational videos and social media campaigns encouraging cancer screening. — Informational videos will be made using community members and will be played in the Blackstone Valley Health Center, as well as posted on social media platforms, such as Facebook and Instagram. These videos will encourage at risk populations in the selected areas to visit their physicians to discuss the possibility of undergoing screening procedures for either breast or colorectal cancer. Data will then be collected about the rates of screening and will be compared to the screening rates from the time period of March 9th 2020 to May 31st 2020, with the goal of increasing screening rates by 25%.

SUMMARY:
Lifespan Cancer Institute serves over 50% of cancer patients in the state. Rhode Island is known for strong medical care and high rates of cancer screening with mammography and colonoscopy. However, cancer screening has plummeted during the COVID-19 pandemic, in part to closing physician offices and stopping non-urgent medical procedures. In addition, anecdotal reports suggest the public remains concerned about returning to physician's offices and risking possible exposure to COVID-19. As in the United States as a whole, COVID-19 has disproportionately impacted ethnic and minority individuals within underserved communities; and in Rhode Island, African Americans, Hispanics and undocumented individuals living in communities such as Central Falls, Pawtucket, Providence, East Providence and North Providence have had the highest rate of COVID-19. These communities are also impacted by healthcare disparities to access and affordability of healthcare, and as such, may be among the least likely to resume cancer screening.

The Lifespan Cancer Institute will institute a project to address health disparities in cancer screening during the pandemic through the use of a targeted campaign involving social media. The goals will be to re-establish screening in the era of COVID-19 and ensure timeliness of care for those found to be at risk, or are positive for, cancer.

DETAILED DESCRIPTION:
This project will focus on improving breast and colorectal cancer screening during the COVID-19 pandemic in underserved populations of Rhode Island. The investigators will engage the Blackstone Valley Community Health Center. Dr. Don Dizon, a national leader in social media, will be a key participant.

Dr. Don Dizon is a world expert using electronic communication and social media in the oncology practice. Dr. Dizon chairs the Digital Engagement Committee for the Southwest Oncology Group (SWOG) a national cancer institute cooperative group. He is a co-principal investigator of an NIH grant studying electronic patient reported outcomes - the SIMPRO Research Consortium. Dr. Dizon is also head of the American Society of Oncology (ASCO) Educational Committee and is well positioned to disseminate the knowledge gathered from the current project through ASCO activities.

The initial project may be to discuss with the Blackstone Valley Community Health Center the possibility of developing short videos in multiple languages on the importance of cancer screening. The investigators will engage staff and patients of the BVCHC and the community to participate within the videos as a model of community-based participation. These informational videos could be distributed directly to the community via social media platforms. Data will be collecting on the rates of cancer screening including age, sex and race. These data could be compared to different cities within Rhode Island and the United States

ELIGIBILITY:
Inclusion Criteria:

* Increased risk of either colorectal or breast cancer
* Living in an under-served area of Rhode Island

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that are at risk of colorectal or breast cancer from under-served or vulnerable communities in Rhode Island.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Increase screening rates for breast and colorectal cancer | 2 years
  Increase screening rates for breast and colorectal cancer among underserved populations by 25% using March 9 through May 31 as a benchmark, coinciding the Executive Orders for COVID19 announced by Governor Raimondo.
Impact of screening on cancer care | 2 years
  Evaluate the impact of screening on timeliness of cancer care among these populations by comparing to the American Society of Clinical Oncology's Quality Oncology Performance Initiative (QOPI) guidelines in breast and colorectal cancer.

SECONDARY OUTCOMES:
Community Engagement | 2 Years
  Evaluate strategies of engagement in these communities as it relates to:
  -Social media platform (Twitter, Facebook, Instagram, TikTok) These metrics will be determined by social media statistics for engagement and the number of calls/queries to the designated information lines.
Barriers to cancer screening during COVID19. | 2 Years
  Evaluate barriers to cancer screening in these populations as it particularly relates to COVID19.

OTHER OUTCOMES:
Educate the community on the importance of cancer screening | 5-10 years
  We will educate staff, community physicians and Rhode Island residents on the importance of cancer screening. We will use community-based partnerships to overcome distrust of institutions and develop an engaged community network. Long term academic goals include publication of data and successfully receiving local and federal funding for continued research.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Lifespan; Don Dizon, MD, Principal Investigator — Lifespan
Locations (1):
- Blackstone Valley Community Health Center, Pawtucket, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- [Background] Wallerstein N, Duran B. Community-based participatory research contributions to intervention research: the intersection of science and practice to improve health equity. Am J Public Health. 2010 Apr 1;100 Suppl 1(Suppl 1):S40-6. doi: 10.2105/AJPH.2009.184036. Epub 2010 Feb 10. PMID 20147663
- [Background] Braun KL, Nguyen TT, Tanjasiri SP, Campbell J, Heiney SP, Brandt HM, Smith SA, Blumenthal DS, Hargreaves M, Coe K, Ma GX, Kenerson D, Patel K, Tsark J, Hebert JR. Operationalization of community-based participatory research principles: assessment of the national cancer institute's community network programs. Am J Public Health. 2012 Jun;102(6):1195-203. doi: 10.2105/AJPH.2011.300304. Epub 2011 Nov 28. PMID 22095340
- [Background] Simonds VW, Wallerstein N, Duran B, Villegas M. Community-based participatory research: its role in future cancer research and public health practice. Prev Chronic Dis. 2013 May 16;10:E78. doi: 10.5888/pcd10.120205. PMID 23680507
- [Background] Alberg AJ, Samet JM. Epidemiology of lung cancer. Chest. 2003 Jan;123(1 Suppl):21S-49S. doi: 10.1378/chest.123.1_suppl.21s. PMID 12527563
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Pham D, Bhandari S, Oechsli M, et al, Lung cancer screening rates: Data from the lung cancer screening registry. J Clin Oncol 36, 2018 (suppl; abstr 6504)
- [Background] Goyal P, Choi JJ, Pinheiro LC, Schenck EJ, Chen R, Jabri A, Satlin MJ, Campion TR Jr, Nahid M, Ringel JB, Hoffman KL, Alshak MN, Li HA, Wehmeyer GT, Rajan M, Reshetnyak E, Hupert N, Horn EM, Martinez FJ, Gulick RM, Safford MM. Clinical Characteristics of Covid-19 in New York City. N Engl J Med. 2020 Jun 11;382(24):2372-2374. doi: 10.1056/NEJMc2010419. Epub 2020 Apr 17. No abstract available. PMID 32302078
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- See also: Blackstone Valley Community Health Center — http://www.bvchc.org/
- See also: Lifespan Cancer Institute — https://www.lifespan.org/centers-services/lifespan-cancer-institute